CLINICAL TRIAL: NCT05893134
Title: Identification of Risk Determinants of Dengue Transmission Through Landscape Analysis in the Neighborhood "El Vergel", Tapachula, Chiapas
Brief Title: Identification of Risk Determinants of Dengue Transmission Through Landscape Analysis
Acronym: IRDDENGUELA
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Instituto Nacional de Salud Publica, Mexico (Other); Centro de Investigación en Matemáticas A.C. (CIMAT) (Unknown)
Responsible Party: Principal Investigator, Héctor Armando Rincón León, Medical Assistant Coordinator for Health Research, State Decentralized Administrative Operation Organ in Chiapas of the Mexican Institute of Social Security, Instituto Mexicano del Seguro Social
Other Study IDs: F-CNIC-2023-060
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Dengue
Keywords: dengue fever; risk determinants; landscape analysis
MeSH Terms: conditions — Dengue | interventions — Risk Assessment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main: Information from entomological, housing condition, and sociodemographic surveys of the El Vergel neighborhood, Tapachula, Chiapas, obtained during the period from November to December 2019, will be used
  Interventions: Other: Risk Assessment

INTERVENTIONS:
Other: Risk Assessment — A probabilistic risk model will be generated based on the variables of different natures used and maps will be built to identify the areas of greatest risk for dengue transmission in the study area

SUMMARY:
This retrospective observational study aims to determine the probability of the risk of dengue transmission through a model based on epidemiological, entomological, socioeconomic, demographic, and landscape variables in the El Vergel neighborhood in the municipality of Tapachula, Chiapas, Mexico.

The main question it aims to answer is:

1. Is it possible to identify the risk determinants of dengue transmission by developing a probabilistic model based on the landscape analysis of epidemiological, entomological, sociodemographic, and landscape variables in an endemic urban area of the municipality of Tapachula, Chiapas, Mexico? Participants will be selected from a registry obtained from the Secretary of Health of cases of dengue fever, which will be contrasted with the entomological, socioeconomic, demographic, and landscape variables in the El Vergel neighborhood in Tapachula, Chiapas, Mexico. They will be not contacted or sampled for biologic testing in any shape or form, only the data already collected from the health services will be used.

DETAILED DESCRIPTION:
Identification of the risk determinants of dengue transmission through landscape analysis in the "El Vergel" neighborhood, Tapachula, Chiapas, Mexico Dengue is a disease transmitted mainly by the Ae. aegypti present in our region, despite vector surveillance and control activities, the circulation of the virus is constant and new strategies are required that contribute to reducing the incidence of the disease, which can be fatal. On the other hand, drones are tools already used in precision and security agriculture, among others; by means of them, it is possible to obtain high-resolution images of large areas of land. This work will use these images in combination with epidemiological, entomological, socioeconomic, and demographic data to identify the risk factors for dengue transmission in an urban area of the city of Tapachula and will generate a model that will allow defining the risk areas in the area. study.

Objective: To determine the probability of the risk of dengue transmission through a model based on epidemiological, entomological, socioeconomic, demographic, and landscape variables in the El Vergel neighborhood in the municipality of Tapachula, Chiapas.

Material and methods: Information from entomological, housing condition, and sociodemographic surveys of the El Vergel neighborhood, Tapachula, Chiapas, obtained during the period from November to December 2019, will be used. In addition to epidemiological information on the incidence of dengue and the placement of ovitraps in the study area during the sampling period, six months before and six months after. Specialized cartography will be used, made from fine-scale aerial photographs taken at a height of 100m by a multirotor drone with six DJI Matrice 600 model rotors with two types of cameras, a Zenmuse X5 model that captures images in the visible spectrum at 16 MP and a multispectral camera with five spectral bands MicaSense RedEdge -MX with RGB sensor with a spatial resolution of 5 cm per pixel. The images were taken simultaneously with the entomological, socioeconomic, and demographic surveys. Georeferenced orthophoto cartographic maps, digital surface models, digital terrain models, and specialized cartography of vegetation indices will be used: Normalized Difference Vegetation Index (NDVI), Difference Vegetation Index Green Normalized (GNDVI), RedEdge Normalized Difference Vegetation Index (NDVIRe) and Chlorophyll Index (CIGreen), height and diameter of the trees present in the study area, to take various variables related to the landscape (environmental variables). The data analysis will be based on a mathematical model based on the principle of partial least squares, to determine the spatial association between the epidemiological indicators (number and georeferencing of cases), entomological (immature and adult stages of Ae. aegypti), condition index housing, sociodemographic and landscape data.

Period: 6 months Type of study: Cross-sectional, retrospective, observational. Selection criteria: The construction of databases will consider the houses of Colonia El Vergel, Tapachula, Chiapas, where its inhabitants of legal age, accepted through informed consent to participate in the surveys and collection of entomological and sociodemographic data in situ and aerial photographs at a height of 100m away. Homes that do not have residents will be grounds for exclusion, and those in which the participants do not allow the collection of complete information will be eliminated.

Sample size and sampling: A multi-stage stratified sampling will be used to select dwellings. The sample size will be obtained according to the sample formula for proportions, which was calculated in n=196 dwellings.

Results: A probabilistic risk model will be generated based on the variables of different natures used and maps will be built to identify the areas of greatest risk for dengue transmission in the study area.

Conclusion: Generate scientific evidence that allows maximum use of these advances for the benefit of populations. The determination of risk areas using specialized cartography carried out using high-resolution aerial photography using drones, has already been demonstrated and recently published.

ELIGIBILITY:
Inclusion Criteria:

* The epidemiological information of all suspected cases of dengue with the onset of symptoms in the period from June 2019 to May 2020 that have a record on the platform of the National System for Epidemiological Surveillance will be included.

Exclusion Criteria:

* Records that do not have sufficient information for their georeferencing will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Health District VII (DSVII) of the State Health Services (SESAs) in Chiapas, Mexico, will be asked for the database of dengue cases in the study area during the time of the implementation of the surveys (November 19 to December 5 of 2019), six months before and six months after the said period. They will be georeferenced through field visits, through the measurement of a geographical point in front of the house.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Risk | One year, six months previous to the survey application (November-December 2019) and six months after
  A probabilistic risk model will be generated based on the variables of different natures used and maps will be built to identify the areas of greatest risk for dengue transmission in the study area

CONTACTS AND LOCATIONS:
Overall Officials: Héctor A Rincón León, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital General de Zona No. 1, Tapachula, Chiapas, Mexico

IPD SHARING:
Plan to Share IPD: No
The information of the participating subjects will only be used for the selection of homes with dengue cases, they will not be contacted or any sample will be obtained, or any drug will be used in them. Therefore, the personal information of the subjects will not be shared in order not to compromise their confidentiality.

REFERENCES:
- [Background] Gubler DJ. Dengue and dengue hemorrhagic fever. Clin Microbiol Rev. 1998 Jul;11(3):480-96. doi: 10.1128/CMR.11.3.480. PMID 9665979
- [Background] Bennett JE, Dolin R, Blaser MJ, editores. Mandell, Douglas, and Bennett's principles and practice of infectious diseases. Ninth edition. Philadelphia, PA: Elsevier; 2020. 1 p.
- [Background] World Health Organization. (2012). Global strategy for dengue prevention and control 2012-2020. World Health Organization. https://apps.who.int/iris/handle/10665/75303
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Brady OJ, Gething PW, Bhatt S, Messina JP, Brownstein JS, Hoen AG, Moyes CL, Farlow AW, Scott TW, Hay SI. Refining the global spatial limits of dengue virus transmission by evidence-based consensus. PLoS Negl Trop Dis. 2012;6(8):e1760. doi: 10.1371/journal.pntd.0001760. Epub 2012 Aug 7. PMID 22880140
- [Background] Kuhn RJ, Zhang W, Rossmann MG, Pletnev SV, Corver J, Lenches E, Jones CT, Mukhopadhyay S, Chipman PR, Strauss EG, Baker TS, Strauss JH. Structure of dengue virus: implications for flavivirus organization, maturation, and fusion. Cell. 2002 Mar 8;108(5):717-25. doi: 10.1016/s0092-8674(02)00660-8. PMID 11893341
- [Background] Guzman MG, Harris E. Dengue. Lancet. 2015 Jan 31;385(9966):453-65. doi: 10.1016/S0140-6736(14)60572-9. Epub 2014 Sep 14. PMID 25230594
- [Background] Pardo Martínez D, Ojeda Martínez B, Alonso Remedios A. Dinámica de la respuesta inmune en la infección por virus del dengue. MediSur. febrero de 2018;16:76-84.
- [Background] Avirutnan P, Matangkasombut P. Unmasking the role of mast cells in dengue. Elife. 2013 Apr 30;2:e00767. doi: 10.7554/eLife.00767. PMID 23638302
- [Background] Orta-Pineda G, Abella-Medrano CA, Suzan G, Serrano-Villagrana A, Ojeda-Flores R. Effects of landscape anthropization on sylvatic mosquito assemblages in a rainforest in Chiapas, Mexico. Acta Trop. 2021 Apr;216:105849. doi: 10.1016/j.actatropica.2021.105849. Epub 2021 Jan 30. PMID 33524383
- [Background] Tun-Lin W, Kay BH, Barnes A. Understanding productivity, a key to Aedes aegypti surveillance. Am J Trop Med Hyg. 1995 Dec;53(6):595-601. doi: 10.4269/ajtmh.1995.53.595. PMID 8561260
- [Background] Scott TW, Morrison AC. Vector dynamics and transmission of dengue virus: implications for dengue surveillance and prevention strategies: vector dynamics and dengue prevention. Curr Top Microbiol Immunol. 2010;338:115-28. doi: 10.1007/978-3-642-02215-9_9. PMID 19802582
- [Background] Reinhold JM, Lazzari CR, Lahondere C. Effects of the Environmental Temperature on Aedes aegypti and Aedes albopictus Mosquitoes: A Review. Insects. 2018 Nov 6;9(4):158. doi: 10.3390/insects9040158. PMID 30404142
- [Background] Carrasco-Escobar G, Moreno M, Fornace K, Herrera-Varela M, Manrique E, Conn JE. The use of drones for mosquito surveillance and control. Parasit Vectors. 2022 Dec 16;15(1):473. doi: 10.1186/s13071-022-05580-5. PMID 36527116
- [Background] Ferraguti M, Martinez-de la Puente J, Roiz D, Ruiz S, Soriguer R, Figuerola J. Effects of landscape anthropization on mosquito community composition and abundance. Sci Rep. 2016 Jul 4;6:29002. doi: 10.1038/srep29002. PMID 27373794
- [Background] Mechan F, Bartonicek Z, Malone D, Lees RS. Unmanned aerial vehicles for surveillance and control of vectors of malaria and other vector-borne diseases. Malar J. 2023 Jan 20;22(1):23. doi: 10.1186/s12936-022-04414-0. PMID 36670398
- [Background] Muñiz-Sánchez, V.; Valdez-Delgado, K.M.; Hernandez-Lopez, F.J.; Moo-Llanes, D.A.; González-Farías, G.; Danis-Lozano, R. Use of Unmanned Aerial Vehicles for Building a House Risk Index of Mosquito-Borne Viral Diseases. Machines 2022, 10, 1161. https://doi.org/10.3390/machines10121161
- [Background] Yin S, Ren C, Shi Y, Hua J, Yuan HY, Tian LW. A Systematic Review on Modeling Methods and Influential Factors for Mapping Dengue-Related Risk in Urban Settings. Int J Environ Res Public Health. 2022 Nov 18;19(22):15265. doi: 10.3390/ijerph192215265. PMID 36429980
- [Background] Leandro AS, Ayala MJC, Lopes RD, Martins CA, Maciel-de-Freitas R, Villela DAM. Entomo-Virological Aedes aegypti Surveillance Applied for Prediction of Dengue Transmission: A Spatio-Temporal Modeling Study. Pathogens. 2022 Dec 20;12(1):4. doi: 10.3390/pathogens12010004. PMID 36678352
- [Background] Hossain, M.S.; Raihan, M.E.; Hossain, M.S.; Syeed, M.M.M.; Rashid, H.; Reza, M.S. Aedes Larva Detection Using Ensemble Learning to Prevent Dengue Endemic. BioMedInformatics 2022, 2, 405-423. https://doi.org/10.3390/biomedinformatics2030026
- [Background] Case E, Shragai T, Harrington L, Ren Y, Morreale S, Erickson D. Evaluation of Unmanned Aerial Vehicles and Neural Networks for Integrated Mosquito Management of Aedes albopictus (Diptera: Culicidae). J Med Entomol. 2020 Sep 7;57(5):1588-1595. doi: 10.1093/jme/tjaa078. PMID 32474595
- [Background] Stanton MC, Kalonde P, Zembere K, Hoek Spaans R, Jones CM. The application of drones for mosquito larval habitat identification in rural environments: a practical approach for malaria control? Malar J. 2021 May 31;20(1):244. doi: 10.1186/s12936-021-03759-2. PMID 34059053
- [Background] Lee GO, Vasco L, Marquez S, Zuniga-Moya JC, Van Engen A, Uruchima J, Ponce P, Cevallos W, Trueba G, Trostle J, Berrocal VJ, Morrison AC, Cevallos V, Mena C, Coloma J, Eisenberg JNS. A dengue outbreak in a rural community in Northern Coastal Ecuador: An analysis using unmanned aerial vehicle mapping. PLoS Negl Trop Dis. 2021 Sep 27;15(9):e0009679. doi: 10.1371/journal.pntd.0009679. eCollection 2021 Sep. PMID 34570788
- [Background] Sallam MF, Fizer C, Pilant AN, Whung PY. Systematic Review: Land Cover, Meteorological, and Socioeconomic Determinants of Aedes Mosquito Habitat for Risk Mapping. Int J Environ Res Public Health. 2017 Oct 16;14(10):1230. doi: 10.3390/ijerph14101230. PMID 29035317
- [Background] Aswi A, Cramb SM, Moraga P, Mengersen K. Bayesian spatial and spatio-temporal approaches to modelling dengue fever: a systematic review. Epidemiol Infect. 2018 Oct 29;147:e33. doi: 10.1017/S0950268818002807. PMID 30369335
- [Background] Rahman MS, Pientong C, Zafar S, Ekalaksananan T, Paul RE, Haque U, Rocklov J, Overgaard HJ. Mapping the spatial distribution of the dengue vector Aedes aegypti and predicting its abundance in northeastern Thailand using machine-learning approach. One Health. 2021 Dec 4;13:100358. doi: 10.1016/j.onehlt.2021.100358. eCollection 2021 Dec. PMID 34934797
- [Background] Abdullah NAMH, Dom NC, Salleh SA, Salim H, Precha N. The association between dengue case and climate: A systematic review and meta-analysis. One Health. 2022 Oct 31;15:100452. doi: 10.1016/j.onehlt.2022.100452. eCollection 2022 Dec. PMID 36561711
- [Background] Talavera JO, Rivas-Ruiz R, Bernal-Rosales LP. [Clinical research V. Sample size]. Rev Med Inst Mex Seguro Soc. 2011 Sep-Oct;49(5):517-22. Spanish. PMID 22185853
- [Background] Moloney JM, Skelly C, Weinstein P, Maguire M, Ritchie S. Domestic Aedes aegypti breeding site surveillance: limitations of remote sensing as a predictive surveillance tool. Am J Trop Med Hyg. 1998 Aug;59(2):261-4. doi: 10.4269/ajtmh.1998.59.261. PMID 9715943
- [Background] Lorenz C, Castro MC, Trindade PMP, Nogueira ML, de Oliveira Lage M, Quintanilha JA, Parra MC, Dibo MR, Favaro EA, Guirado MM, Chiaravalloti-Neto F. Predicting Aedes aegypti infestation using landscape and thermal features. Sci Rep. 2020 Dec 10;10(1):21688. doi: 10.1038/s41598-020-78755-8. PMID 33303912
- [Background] Arredondo-Jimenez JI, Valdez-Delgado KM. Aedes aegypti pupal/demographic surveys in southern Mexico: consistency and practicality. Ann Trop Med Parasitol. 2006 Apr;100 Suppl 1:S17-S32. doi: 10.1179/136485906X105480. PMID 16630388
- [Background] Silver JB. Mosquito ecology: field sampling methods. springer science & business media; 2007.
- [Result] Valdez-Delgado KM, Moo-Llanes DA, Danis-Lozano R, Cisneros-Vazquez LA, Flores-Suarez AE, Ponce-Garcia G, Medina-De la Garza CE, Diaz-Gonzalez EE, Fernandez-Salas I. Field Effectiveness of Drones to Identify Potential Aedes aegypti Breeding Sites in Household Environments from Tapachula, a Dengue-Endemic City in Southern Mexico. Insects. 2021 Jul 21;12(8):663. doi: 10.3390/insects12080663. PMID 34442229
- [Result] Valdez-Delgado KM. Aplicación del uso de drones a fina escala para la asociación de factores demográficos, socio-económicos y ambientales con la abundancia de mosquitos Aedes aegypti (Linnaeus) y Aedes albopictus (Skuse) Diptera: Culicidae, en áreas persistentes para la transmisión de dengue, chikungunya y Zika de la Ciudad de Tapachula, Chiapas". [Internet] [Tesis Doctoral]. [Monterrey, NL]: Universidad Autónoma de Nuevo León; 2023. Disponible en: http://eprints.uanl.mx/id/eprint/25097